CLINICAL TRIAL: NCT00215332
Title: Five-year Follow-up of the CHARITÉ™ Artificial Disc Compared to Anterior Lumbar Interbody Fusion With the BAK Cage.
Brief Title: CHARITE™ vs. ALIF 5-Year Follow-up
Status: Completed | Type: Observational
Sponsor: DePuy Spine (Industry)
Other Study IDs: P040006
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Degenerative Disc Disease
Keywords: arthroplasty; lumbar; disc
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Training- CHARITE: Non-Randomized Training (TDR with CHARITE)
  Interventions: Device: CHARITE
- CHARITE: Randomized Subjects treated by Lumbar Total Disc Replacment with CHARITE
  Interventions: Device: CHARITE
- Control: Randomized Subjects treated by ALIF with BAK cage

INTERVENTIONS:
Device: CHARITE — Lumbar Total Disc Replacement
  Groups: CHARITE; Training- CHARITE

SUMMARY:
To assess the clinical and radiographic outcomes through 5-years following treatment with CHARITÉ™ Artificial Disc vs. the BAK Cage for treatment of degenerative disc disease at one level (L4-S1).

DETAILED DESCRIPTION:
This study is an extension out to 5 year follow-up of a randomized comparative IDE trial of the CHARITÉ™ Artificial Disc vs. ALIF with the BAK cage for treatment of degenerative disc disease. The original 2-year trial demonstrated non-inferiority of the CHARITÉ™ compared to ALIF.

This extension will continue to follow-up the original outcome measures and will also examine adjacent segment progression.

ELIGIBILITY:
Inclusion Criteria:

* Participated in either the training or randomized arm of the CHARITÉ Artificial Disc IDE study,
* Still have the original implant they received in their index surgery.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 367 (Estimated)
Dates: Start 2005-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall Success | 5 Years
  ODI Improvement greater than or equal to 15 points from baseline No device failures (i.e., revision, re-operation, supplemental fixation, or removal) No major complications Maintenance or improvement in neurological status compared to baseline.

SECONDARY OUTCOMES:
Secondary Endpoints | 5 Years
  Components of the Overall Success definition (neurological and ODI scores) Visual Analog Scale (VAS) Disc height Range of Motion Migration of the device Radiolucency

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Stoutenburgh, Study Director — DePuy Spine
Locations (10):
- United States (10):
  - Charite Site 13, Los Angeles, California
  - Charite Site 06, Golden, Colorado
  - Charite Site 11, Chicago, Illinois
  - Charite Site 03, Louisville, Kentucky
  - Charite Site 02, Towson, Maryland
  - Charite Site 15, Boston, Massachusetts
  - Charite Site 14, Lockport, New York
  - Charite Site 10, New York, New York
  - Charite Site 07, Columbus, Ohio
  - Charite Site 01, Plano, Texas